CLINICAL TRIAL: NCT06691659
Title: Next-Generation Photon-Counting CT Technology: Development and Clinical Evaluation
Acronym: CT-DACE
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Canon Medical Systems, USA (Industry)
Responsible Party: Sponsor
Other Study IDs: 856690
Record Dates: First submitted 2024-11-11; First posted 2024-11-15 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Radiation Protection; Image Enhancement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT-DACE — Photon Counting CT scan

SUMMARY:
This project aims to develop and evaluate a next-generation photon-counting CT prototype, and assess whether next-generation photon-counting CT--which enables reduced radiation dose, high spatial resolution, and spectral imaging--would facilitate improved diagnostic performance for abdominal, cardiothoracic, musculoskeletal, and neuroimaging.

DETAILED DESCRIPTION:
This protocol aims to assess the diagnostic benefits of a next-generation Photon-Counting Computed Tomography (PCCT) system in patients undergoing routine CT imaging.

Recruitment will be conducted among patients scheduled for CT scans (with or without contrast agent) at the Perelman Center for Advanced Medicine. Patients in the study will undergo abdominal, cardiovascular, chest, musculoskeletal, and neuroimaging scans.

The design involves 50 participants per body region to gather preliminary data and assess diagnostic benefits for future research and clinical translation.

This a total of 250 patients for the initial study.

Analyses will be conducted as needed, based on the specific validation or quantitative measures required for each clinical CT scan. This study will involve three radiologists for each cohort, selected based on their training in the specific anatomical region of interest, analyzing images from PCCT scanning. They will interpret both conventional CT slices and the additional spectral and high-resolution data provided by the PCCT. The images will be reviewed on a state-of-the-art workstation with a high-resolution monitor. Performance metrics will be set individually for each anatomical region.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 89.
* Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.
* Not pregnant (based on attestation)

Exclusion Criteria:

* Pregnant women will not be included. All females of childbearing potential must attest that they are not pregnant before CT imaging.
* Participants with a known contrast allergy.
* Any current medical condition, illness, or disorder, as assessed by medical record review and/or self-reported, that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study.

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Recruited patients are scheduled to undergo a routine CT scan (with or without contrast) at the Perelman Center for Advanced Medicine.
  Patients in the study will undergo abdominal, cardiovascular, chest, musculoskeletal, and neuroimaging scans. The design involves 50 participants per body region to gather preliminary data and assess diagnostic benefits for future research and clinical translation.
  This a total of 250 patients for the initial study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 24 months
  In this clinical study evaluating a photon-counting computed tomography (CT) scanner, the Primary Outcome Measures include image quality assessed by signal-to-noise ratio, contrast-to-noise ratio, and resolution via edge response function, as well as diagnostic accuracy determined by radiologist interpretation compared to gold-standard diagnostic methods when available from previous scans.
  For each body region, image data will be subjectively evaluated for image quality using a Likert scale assessing overall image quality, presence of artifacts, and diagnostic adequacy for the specific clinical indication.

CONTACTS AND LOCATIONS:
Overall Officials: Peter B Noel, PhD, Principal Investigator — UPENN Radiology
Locations (1):
- University of Pennsylvania - Center for Advanced Computed Tomography Imaging Services (CACTIS), Philadelphia, Pennsylvania, United States